CLINICAL TRIAL: NCT06518044
Title: N-acetyl-L-cysteine for Promoting Hematopoietic Recovery in Patients With Severe Aplastic Anemia (SAA) After Haploidentical Transplantation -- a Prospective Single-arm Clinical Study
Brief Title: NAC for Hematopoietic Recovery in SAA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAC in SAA post haplo-HSCT
Record Dates: First submitted 2024-06-29; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Aplastic Anemia
Keywords: hematopoietic recovery; NAC; HSCT
MeSH Terms: conditions — Anemia, Aplastic | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NAC group (Experimental): Aplastic anemia patients receiving haploidentical transplantation will be enrolled, and NAC (400mg tid) will be administered orally from day 14 before conditioning until day +60 post-HSCT. The initial dose of NAC was 400mg orally three times daily (TID).
  Interventions: Drug: N Acetyl L Cysteine

INTERVENTIONS:
Drug: N Acetyl L Cysteine — For subjects in the experimental intervention arm (NAC group), if the patients met the inclusion criteria on day 14 before conditioning, they received NAC from day 14 before conditioning until day +60 post-HSCT. The initial dose of NAC was 400mg orally three times daily (TID). In cases of grade 3 or worse AEs (not including hematologic recovery), dose modifications including dose reductions or interruptions were permitted at the physician's discretion. After the resolution of AEs, the dose was re-escalated from to 400mg TID.

SUMMARY:
This is a prospective single-arm clinical study to evaluate the role of NAC among patients with severe aplastic anemia (SAA) can promote hematopoietic recovery after haploidentical transplantation.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective treatment of severe aplastic anemia (SAA). However, poor hematopoietic reconstitution including poor graft function (PGF) and prolonged isolated thrombocytopenia (PT), remains a life-threatening complication after allo-HSCT. Especially with the increasing use of haploidentical allo-HSCT (haplo-HSCT) in the past ten years, PGF and PT have become growing obstacles contributing to high morbidity and mortality after allo-HSCT. A previous clinical prospective cohort study showed that NAC could improve the function of bone marrow endothelial progenitor cells and promote hematopoietic recovery among leukemia patients after haploidentical transplantation. Therefore, we hypothesized that the prophylactic administration of NAC could facilitate the recovery of hematopoietic capacity by improving the bone marrow microenvironment of patients with SAA after haploidentical transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with SAA or vSAA
2. Aged 18-50
3. No severe organ injury
4. No uncontrolled active infections
5. Sign informed consent form, have the ability to comply with study and follow-up procedures

Exclusion Criteria:

1. Hypersensitivity to NAC or history of bronchial asthma
2. Life expectancy less than 30 days post-transplantation
3. Uncontrolled infections pre-transplantation
4. Cardiac dysfunction (particularly congestive heart failure, unstable coronary artery disease and serious cardiac ventricular arrhythmias requiring antiarrhythmic therapy)
5. Respiratory failure ( PaO2 ≤60mmHg)
6. Hepatic abnormalities (total bilirubin ≥2 times the upper limit of normal [ULN], alanine aminotransferase or aspartate aminotransferase ≥2 times the ULN)
7. Renal dysfunction (creatinine ≥1.5 times the ULN or creatinine clearance rate < 30 mL/min)
8. ECOG performance status ≥3
9. With any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of prolonged thrombcytopenia (PT), which was assessed at +2M post-HSCT. | Two months post-HSCT.
  PT was defined as platelet count less than 20×109/L or a dependence on platelet transfusion with the engraftment of other cell lines(ANC>0.5×109/L and hemoglobin>70 g/L without transfusion support) beyond day +60 post-HSCT in the presence of complete donor chimerism (CDC).
The incidence of poor graft function (PGF), which was assessed at +2M post-HSCT. | Two months post-HSCT.
  PGF was defined as the presence of 2 or 3 cytopenic counts (ANC≤0.5×109/L, platelet≤20×109/L, or hemoglobin≤70 g/L) for at least 3 consecutive days beyond day +28 post-HSCT with a transfusion requirement, related with hypoplastic-aplastic BM, in the presence of complete donor chimerism (CDC).

SECONDARY OUTCOMES:
The cumulative incidences of transplantation related mortality (TRM). | Two months post-HSCT.
  Number of participants suffered TRM will be calculated.
The cumulative incidences of Thrombotic Microangiopathy (TMA). | Two months post-HSCT.
  Number of participants suffered TMA will be calculated.
The cumulative incidences of graft versus host disease (GvHD). | Two months post-HSCT.
  Number of participants suffered GvHD will be calculated.
The cumulative incidences of overall survival (OS). | One year post-HSCT.
  Number of participants survived for 1 year post diagnosed will be calculated.
Adverse reactions | Two months post-HSCT.
  Liver function, renal function, respiratory syndrom assessed by CTCAE v4.0 during oral administration of NAC.

IPD SHARING:
Plan to Share IPD: No